CLINICAL TRIAL: NCT01248884
Title: Safety and Immunogenicity of New Formulations of GlaxoSmithKline Biologicals' DTPa-HBV-IPV/Hib Vaccine (GSK217744) in Primary Infant Vaccination
Brief Title: Safety and Immunogenicity of New Formulations of GlaxoSmithKline Biologicals' DTPa-HBV-IPV/Hib Vaccine (GSK217744)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 113948
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2014-07

CONDITIONS: Tetanus; Poliomyelitis; Hepatitis B; Haemophilus Influenzae Type b; Acellular Pertussis; Diphtheria
Keywords: combination vaccine; Primary vaccination
MeSH Terms: conditions — Tetanus; Poliomyelitis; Hepatitis B; Haemophilus Infections; Diphtheria | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- GSK217744 Group 1 (Experimental): Subjects aged between and including 60 and 90 days of age at the time of first vaccination received 3 doses of GSK217744 formulation A vaccine, co-administered with Prevenar 13® at 2, 3 and 4 months of age. The GSK217744 and Prevenar 13® vaccines were administered intramuscularly into the left and right sides of the thigh, respectively.
  Interventions: Biological: Prevenar 13®; Biological: GSK217744
- GSK217744 Group 2 (Experimental): Subjects aged between and including 60 and 90 days of age at the time of first vaccination received 3 doses of GSK217744 formulation B vaccine, co-administered with Prevenar 13® at 2, 3 and 4 months of age. The GSK217744 and Prevenar 13® vaccines were administered intramuscularly into the left and right sides of the thigh, respectively.
  Interventions: Biological: Prevenar 13®; Biological: GSK217744
- Infanrix hexa Group (Active Comparator): Subjects aged between and including 60 and 90 days of age at the time of first vaccination received 3 doses of Infanrix hexa™ vaccine, co-administered with Prevenar 13® at 2, 3 and 4 months of age. The Infanrix hexa™ and Prevenar 13® vaccines were administered intramuscularly into the left and right sides of the thigh, respectively.
  Interventions: Biological: Infanrix hexa™; Biological: Prevenar 13®

INTERVENTIONS:
Biological: Infanrix hexa™ — 3 doses, intramuscular into left thigh
  Other Names: DTPa-HBV-IPV/Hib
  Arms: Infanrix hexa Group
Biological: Prevenar 13® — 3 co-administered doses, intramuscular into right thigh
  Other Names: Pfizer's 13-valent pneumococcal polysaccharide conjugate vaccine
Biological: GSK217744 — 3 doses, intramuscular into left thigh
  Arms: GSK217744 Group 1; GSK217744 Group 2

SUMMARY:
This study is designed to evaluate the safety and immunogenicity of new formulations of GSK Biologicals' DTPa-HBV-IPV/Hib vaccine (GSK217744) when administered as a primary vaccination course to healthy infants at 2, 3 and 4 months of age.

DETAILED DESCRIPTION:
This Protocol Posting has been updated following Protocol Amendment 1, February 2011, leading to the update of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between, and including, 60 and 90 days of age at the time of the first vaccination.
* Born after a gestation period of 37 to 42 weeks inclusive.
* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/ Legally Acceptable Representative(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Administration of a vaccine not foreseen by the study protocol, within 30 days prior to the first study visit, or planned administration during the study period, with the exception of oral rotavirus vaccination which is allowed at any time during the study.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Evidence of previous or intercurrent diphtheria, tetanus, pertussis, polio, hepatitis B, Hib and/or pneumococcal vaccination or disease, with the exception of hepatitis B vaccination at birth.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Acute disease and/or fever at the time of enrolment.

Ages: 60 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 721 (Actual)
Dates: Start 2010-12-09; Primary Completion 2012-01-05 (Actual); Study Completion 2012-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- Dominican Republic (2):
  - GSK Investigational Site, Santo Domingo
  - GSK Investigational Site, Santo Domingo, Distrito Nacional
- Finland (12):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa

REFERENCES:
- [Derived] Vesikari T, Rivera L, Korhonen T, Ahonen A, Cheuvart B, Hezareh M, Janssens W, Mesaros N. Immunogenicity and safety of primary and booster vaccination with 2 investigational formulations of diphtheria, tetanus and Haemophilus influenzae type b antigens in a hexavalent DTPa-HBV-IPV/Hib combination vaccine in comparison with the licensed Infanrix hexa. Hum Vaccin Immunother. 2017 Jul 3;13(7):1505-1515. doi: 10.1080/21645515.2017.1294294. Epub 2017 Mar 24. PMID 28340322

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 721 subjects were enrolled in the study.
Groups:
- Infanrix Hexa Group: Subjects aged between and including 60 and 90 days of age at the time of first vaccination received 3 doses of Infanrix hexa™ vaccine, co-administered with Prevenar 13® at 2, 3 and 4 months of age. The Infanrix hexa™ and Prevenar 13® vaccines were administered intramuscularly into the left and right sides of the thigh, respectively .
Period: Overall Study
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Started | 240 | 242 | 239
Completed | 238 | 239 | 238
Not Completed | 2 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 1
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group | Total
Number analyzed (Participants) | 240 | 242 | 239 | 721
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 9.7 (1.36) | 9.8 (1.29) | 9.7 (1.21) | 9.73 (1.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 138 | 99 | 356
  Male | 121 | 104 | 140 | 365
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage /African American | 1 | 0 | 1 | 2
  White - Arabic / north African heritage | 3 | 1 | 6 | 10
  White - Caucasian / European heritage | 144 | 148 | 140 | 432
  Unspecified | 92 | 93 | 92 | 277

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects for Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies.
Description: A seroprotected subject was defined as a vaccinated subject who had anti-D and anti-T antibody concentrations ≥ 0.1 international units per milliliter (IU/mL).
Time Frame: At Month 0
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects, who complied with the protocol, for whom immunogenicity data were available and for whom assay results were available for antibodies against at least one study vaccine antigen component after at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 200 | 210 | 211
Participants
  Anti-D | 154 | 165 | 160
  Anti-T | 197 | 206 | 209

2. Primary Outcome: Number of Seroprotected Subjects for Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies.
Description: as for outcome 1
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 214 | 217 | 219
Participants
  Anti-D | 214 | 217 | 219
  Anti-T | 214 | 217 | 219
Statistical Analysis 1: Comparison: GSK217744 Group 1 vs Infanrix Hexa Group; Test type: Non-Inferiority — Non-inferiority in terms of immune response to diphteria antigens was demonstrated if the upper limit of the 97.5% confidence interval (CI) on the group difference (Infanrix hexa Group minus GSK2177744 Group 1) in the percentage of seroprotected subject was below or equal to 10%; Difference in percentage = 0, 97.5% CI 2-sided [-2.25 to 2.3]
Statistical Analysis 2: Comparison: GSK217744 Group 1 vs Infanrix Hexa Group; Test type: Non-Inferiority — Non-inferiority in terms of immune response to tetanus antigens was demonstrated if the upper limit of the 97.5% confidence interval (CI) on the group difference (Infanrix hexa Group minus GSK2177744 Group 1) in the percentage of seroprotected subject was below or equal to 10%; Difference in percentage = 0, 97.5% CI 2-sided [-2.25 to 2.3]
Statistical Analysis 3: Comparison: GSK217744 Group 2 vs Infanrix Hexa Group; Test type: Non-Inferiority — Non-inferiority in terms of immune response to diphteria antigens was demonstrated if the upper limit of the 97.5% confidence interval (CI) on the group difference (Infanrix hexa Group minus GSK2177744 Group 2) in the percentage of seroprotected subject was below or equal to 10%; Difference in percentage = 0, 97.5% CI 2-sided [-2.25 to 2.27]
Statistical Analysis 4: Comparison: GSK217744 Group 2 vs Infanrix Hexa Group; Test type: Non-Inferiority — Non-inferiority in terms of immune response to tetanus antigens was demonstrated if the upper limit of the 97.5% confidence interval (CI) on the group difference (Infanrix hexa Group minus GSK2177744 Group 2) in the percentage of seroprotected subject was below or equal to 10%; Difference in percentage = 0, 97.5% CI 2-sided [-2.25 to 2.27]

3. Primary Outcome: Concentrations for Anti-pertussis Toxoid (Anti-PT) and Anti-pertactin (Anti-PRN) Antibodies.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seroprotection cut-off of the assay was ≥ 5 enzyme-linked immunosorbent assay (ELISA) units per milliliters (EL.U/mL).
Time Frame: At Month 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 200 | 210 | 210
EL.U/mL
  Anti-PT: number analyzed (Participants) | 199 | 210 | 210
  Anti-PT | 3.3 [3.0 to 3.6] | 3.4 [3.1 to 3.7] | 3.1 [2.9 to 3.4]
  Anti-PRN | 5.1 [4.5 to 5.9] | 4.9 [4.3 to 5.5] | 4.9 [4.3 to 5.7]

4. Primary Outcome: Concentrations for Anti-pertussis Toxoid (Anti-PT) and Anti-pertactin (Anti-PRN) Antibodies.
Description: as for outcome 3
Time Frame: At Month 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 215 | 217 | 219
EL.U/mL
  Anti-PT: number analyzed (Participants) | 215 | 217 | 218
  Anti-PT | 57.7 [52.9 to 62.9] | 57.5 [53.1 to 62.4] | 73.2 [67.7 to 79.2]
  Anti-PRN: number analyzed (Participants) | 214 | 215 | 219
  Anti-PRN | 76.6 [68.1 to 86.3] | 65.7 [58.9 to 73.3] | 106.6 [96.6 to 117.8]
Statistical Analysis 1: Comparison: GSK217744 Group 1 vs Infanrix Hexa Group; Test type: Non-Inferiority — Non-inferiority in terms of immune response to pertussis antigen (anti-PT) was demonstrated if the upper limit of the 97.5% confidence interval (CI) on the GMC ratio (Infanrix hexa Group divided by GSK2177744 Group 1) was below or equal to 1.5; GMC ratio = 1.26, 97.5% CI 2-sided [1.11 to 1.44]
Statistical Analysis 2: Comparison: GSK217744 Group 1 vs Infanrix Hexa Group; Test type: Non-Inferiority — Non-inferiority in terms of immune response to pertussis antigen (anti-PRN) was demonstrated if the upper limit of the 97.5% confidence interval (CI) on the GMC ratio (Infanrix hexa Group divided by GSK2177744 Group 1) was below or equal to 1.5; GMC ratio = 1.33, 97.5% CI 2-sided [1.14 to 1.54]
Statistical Analysis 3: Comparison: GSK217744 Group 2 vs Infanrix Hexa Group; Test type: Non-Inferiority — Non-inferiority in terms of immune response to pertussis antigen (anti-PT) was demonstrated if the upper limit of the 97.5% confidence interval (CI) on the GMC ratio (Infanrix hexa Group divided by GSK2177744 Group 2) was below or equal to 1.5; GMC ratio = 1.25, 97.5% CI 2-sided [1.1 to 1.43]
Statistical Analysis 4: Comparison: GSK217744 Group 2 vs Infanrix Hexa Group; Test type: Non-Inferiority — Non-inferiority in terms of immune response to pertussis antigen (anti-PRN) was demonstrated if the upper limit of the 97.5% confidence interval (CI) on the GMC ratio (Infanrix hexa Group divided by GSK2177744 Group 2) was below or equal to 1.5; GMC ratio = 1.58, 97.5% CI 2-sided [1.37 to 1.84]

5. Primary Outcome: Number of Seroprotected Subjects for Anti-polyribosyl-ribitol-phosphate (Anti-PRP) Antibodies.
Description: A seroprotected subject was defined as a vaccinated subject who had anti-PRP antibody concentrations ≥ 0.15 micrograms per milliliter (µg/mL).
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 214 | 216 | 218
Participants | 197 | 190 | 193
Statistical Analysis 1: Comparison: GSK217744 Group 1 vs Infanrix Hexa Group; Test type: Non-Inferiority — Non-inferiority in terms of immune response to PRP antigens was demonstrated if the upper limit of the 97.5 confidence interval (CI) on the group difference (Infanrix hexa Group minus GSK217744 Group 1) in the percentage of seroprotected subjects was below or equal to 10%; Difference in percentage = -3.52, 97.5% CI 2-sided [-10.19 to 3]
Statistical Analysis 2: Comparison: GSK217744 Group 2 vs Infanrix Hexa Group; Test type: Non-Inferiority — Non-inferiority in terms of immune response to PRP antigens was demonstrated if the upper limit of the 97.5 confidence interval (CI) on the group difference (Infanrix hexa Group minus GSK217744 Group 2) in the percentage of seroprotected subjects was below or equal to 10%; Difference in percentage = 0.57, 97.5% CI 2-sided [-6.53 to 7.7]

6. Primary Outcome: Number of Subjects With Anti-hepatitis B (Anti-HBs) Antibody Concentration Equal to or Above (≥) 10 and 100 Milli-International Units Per Milliliter (mIU/mL)
Description: A seroprotected subject was defined as a vaccinated subject who had anti-HBs antibody concentrations ≥ 10 mIU/mL. A decrease in the specificity of the anti-HB enzyme-linked immunosorbent assay (ELISA) had been observed in some studies for low levels of antibody (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Infanrix Hexa Group: Subjects aged between and including 60 and 90 days of age at the time of first vaccination received 3 doses of Infanrix hexaTM vaccine, co-administered with Prevenar 13® at 2, 3 and 4 months of age. The Infanrix hexaTM and Prevenar 13® vaccines were administered intramuscularly into the left and right sides of the thigh, respectively.
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 202 | 205 | 209
Participants
  Anti-HBs ≥ 10 mIU/mL (ELISA) | 197 | 203 | 205
  Anti-HBs ≥ 100 mIU/mL (ELISA) | 184 | 183 | 196
  Anti-HBs ≥ 10 mIU/mL (CLIA) | 197 | 201 | 203
Statistical Analysis 1: Comparison: GSK217744 Group 1 vs Infanrix Hexa Group; Immune response non-inferiority - anti-HBs (ELISA); Test type: Non-Inferiority — Non-inferiority in terms of immune response to hepatitis B (HBs) antigens was demonstrated if the upper limit of the 97.5 confidence interval (CI) on the group difference (Infanrix hexa minus GSK217744 Group 1) in the percentage of seroprotected subjects was below or equal to 10%; Difference in percentage = 0.56, 97.5% CI 2-sided [-3.27 to 4.63]
Statistical Analysis 2: Comparison: GSK217744 Group 2 vs Infanrix Hexa Group; Immune response non-inferiority - anti-HBs (ELISA); Test type: Non-Inferiority — Non-inferiority in terms of immune response to hepatitis B (HBs) antigens was demonstrated if the upper limit of the 97.5 confidence interval (CI) on the group difference (Infanrix hexa minus GSK217744 Group 2) in the percentage of seroprotected subjects was below or equal to 10%; Difference in percentage = -0.94, 97.5% CI 2-sided [-4.57 to 2.36]
Statistical Analysis 3: Comparison: GSK217744 Group 1 vs Infanrix Hexa Group; Immune response non-inferiority - anti-HBs (CLIA); Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Difference in percentage = -0.4, 97.5% CI 2-sided [-4.62 to 3.8]
Statistical Analysis 4: Comparison: GSK217744 Group 2 vs Infanrix Hexa Group; Immune response non-inferiority - anti-HBs (CLIA); Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Difference in percentage = -0.92, 97.5% CI 2-sided [-5.07 to 3.02]

7. Primary Outcome: Concentrations for Anti-HBs Antibodies ≥ 10 and 100 mIU/mL
Description: A decrease in the specificity of the anti-HB enzyme-linked immunosorbent assay (ELISA) had been observed in some studies for low levels of antibody (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis. Concentrations were expressed as geometric mean concentrations (GMCs) in milli-International units per milliliter (mIU/mL).
Time Frame: At Month 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 202 | 205 | 209
mIU/mL | 639.5 [523.6 to 781.2] | 602.6 [492.1 to 737.9] | 799.0 [662.2 to 964.0]

8. Secondary Outcome: Concentrations for Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seroprotection cut-off of the assay was 0.1 IU/mL.
Time Frame: At Months 0 and 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 214 | 217 | 219
IU/mL
  Anti-D at Month 0: number analyzed (Participants) | 200 | 210 | 211
  Anti-D at Month 0 | 0.292 [0.247 to 0.347] | 0.281 [0.238 to 0.332] | 0.290 [0.245 to 0.343]
  Anti-D at Month 3 | 1.499 [1.367 to 1.644] | 1.704 [1.564 to 1.856] | 1.839 [1.686 to 2.005]
  Anti-T at Month 0: number analyzed (Participants) | 200 | 210 | 211
  Anti-T at Month 0 | 0.936 [0.832 to 1.053] | 0.920 [0.822 to 1.029] | 0.907 [0.812 to 1.013]
  Anti-T at Month 3 | 1.761 [1.624 to 1.910] | 1.726 [1.597 to 1.865] | 1.947 [1.818 to 2.085]

9. Secondary Outcome: Number of Seropositive Subjects for Anti-pertussis Toxoid (Anti-PT) and Anti-pertactin (Anti-PRN) Antibodies.
Description: A seropositive subject was defined as a vaccinated subject who had anti-PT and anti-PRN antibody concentrations ≥ 5 EL.U/mL.
Time Frame: At Months 0 and 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 215 | 217 | 219
Participants
  Anti-PT at Month 0: number analyzed (Participants) | 199 | 210 | 210
  Anti-PT at Month 0 | 33 | 38 | 31
  Anti-PT at Month 3: number analyzed (Participants) | 215 | 217 | 218
  Anti-PT at Month 3 | 215 | 217 | 218
  Anti-PRN at Month 0: number analyzed (Participants) | 200 | 210 | 210
  Anti-PRN at Month 0 | 84 | 89 | 76
  Anti-PRN at Month 3: number analyzed (Participants) | 214 | 215 | 219
  Anti-PRN at Month 3 | 214 | 215 | 219

10. Secondary Outcome: Concentrations for Anti-polyribosyl-ribitol-phosphate (Anti-PRP) Antibodies.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seroprotection cut-off of the assay was ≥ 0.15 µg/mL.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 214 | 216 | 218
µg/mL | 0.951 [0.793 to 1.142] | 0.730 [0.606 to 0.880] | 1.082 [0.884 to 1.324]

11. Secondary Outcome: Number of Seropositive Subjects for Anti-pneumococcal (Anti-PNE) Serotypes.
Description: A seropositive subject was defined as a vaccinated subject who had anti- pneumococcal antibody concentrations ≥ 0.15 micrograms per milliliter (µg/mL). The anti-PNE serotypes assessed were 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 108 | 112 | 114
Participants
  Anti- PNE 1: number analyzed (Participants) | 107 | 112 | 112
  Anti- PNE 1 | 107 | 112 | 111
  Anti- PNE 3: number analyzed (Participants) | 106 | 105 | 107
  Anti- PNE 3 | 106 | 105 | 107
  Anti- PNE 4 | 108 | 112 | 114
  Anti- PNE 5: number analyzed (Participants) | 108 | 111 | 112
  Anti- PNE 5 | 107 | 109 | 109
  Anti- PNE 6A | 108 | 111 | 112
  Anti- PNE 6B: number analyzed (Participants) | 107 | 112 | 113
  Anti- PNE 6B | 97 | 104 | 102
  Anti- PNE 7F | 107 | 111 | 114
  Anti- PNE 9V | 107 | 112 | 113
  Anti- PNE 14 | 108 | 112 | 114
  Anti- PNE 18C: number analyzed (Participants) | 108 | 112 | 113
  Anti- PNE 18C | 106 | 112 | 109
  Anti- PNE 19A: number analyzed (Participants) | 106 | 112 | 114
  Anti- PNE 19A | 106 | 112 | 114
  Anti- PNE 19F | 107 | 111 | 114
  Anti- PNE 23F | 103 | 104 | 108

12. Secondary Outcome: Concentrations for Anti-PNE Antibodies.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seropositivity cut-off of the assay was 0.15 µg /mL. The anti-PNE serotypes assessed were 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg /mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 108 | 112 | 114
µg /mL
  Anti- PNE 1: number analyzed (Participants) | 107 | 112 | 112
  Anti- PNE 1 | 1.61 [1.42 to 1.83] | 1.48 [1.32 to 1.67] | 1.58 [1.38 to 1.81]
  Anti- PNE 3: number analyzed (Participants) | 106 | 105 | 107
  Anti- PNE 3 | 0.91 [0.80 to 1.03] | 0.91 [0.82 to 1.01] | 0.94 [0.84 to 1.05]
  Anti- PNE 4 | 1.80 [1.61 to 2.03] | 1.62 [1.47 to 1.80] | 1.69 [1.50 to 1.90]
  Anti- PNE 5: number analyzed (Participants) | 108 | 111 | 112
  Anti- PNE 5 | 0.79 [0.69 to 0.89] | 0.77 [0.69 to 0.87] | 0.82 [0.72 to 0.93]
  Anti- PNE 6A | 1.63 [1.39 to 1.91] | 1.43 [1.23 to 1.66] | 1.52 [1.30 to 1.79]
  Anti- PNE 6B: number analyzed (Participants) | 107 | 112 | 113
  Anti- PNE 6B | 0.66 [0.53 to 0.82] | 0.64 [0.52 to 0.78] | 0.69 [0.56 to 0.85]
  Anti- PNE 7F | 2.18 [1.91 to 2.49] | 2.30 [2.05 to 2.59] | 2.48 [2.20 to 2.79]
  Anti- PNE 9V | 1.12 [0.97 to 1.28] | 1.11 [0.99 to 1.25] | 1.16 [1.02 to 1.32]
  Anti- PNE 14 | 7.47 [6.33 to 8.81] | 7.80 [6.79 to 8.96] | 8.03 [6.81 to 9.48]
  Anti- PNE 18C: number analyzed (Participants) | 108 | 112 | 113
  Anti- PNE 18C | 1.56 [1.33 to 1.84] | 1.55 [1.39 to 1.74] | 1.56 [1.33 to 1.82]
  Anti- PNE 19A: number analyzed (Participants) | 106 | 112 | 114
  Anti- PNE 19A | 2.70 [2.35 to 3.09] | 2.75 [2.40 to 3.15] | 2.68 [2.38 to 3.03]
  Anti- PNE 19F | 2.55 [2.16 to 3.00] | 2.53 [2.19 to 2.92] | 2.79 [2.44 to 3.18]
  Anti- PNE 23F | 0.89 [0.73 to 1.09] | 0.83 [0.69 to 1.01] | 0.91 [0.75 to 1.10]

13. Secondary Outcome: Number of Subjects With a Vaccine Response to PT and PRN.
Description: Vaccine response defined as: for initially seronegative subjects, antibody concentration ≥ 5 EL.U/mL at 1 month post primary vaccination (Month 3); for initially seropositive subjects, antibody concentration at 1 month post primary vaccination (Month 3) ≥ 1 fold the pre-vaccination antibody concentration.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 199 | 210 | 210
Participants
  Anti- PT: number analyzed (Participants) | 199 | 210 | 209
  Anti- PT | 195 | 204 | 207
  Anti- PRN: number analyzed (Participants) | 199 | 208 | 210
  Anti- PRN | 181 | 194 | 198

14. Secondary Outcome: Number of Subjects Reporting Any Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of any local symptom regardless of intensity grade.
Time Frame: During the 8-day (Days 0-7)
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 240 | 240 | 238
Participants
  Any pain | 190 | 183 | 155
  Any redness | 151 | 140 | 128
  Any swelling | 124 | 122 | 115

15. Secondary Outcome: Number of Subjects Reporting Any Solicited General Symptoms.
Description: Solicited local symptoms assessed were drowsiness, irritability, loss of appetite and fever [axillary temperature above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of any local symptom regardless of intensity grade.
Time Frame: During the 8-day (Days 0-7)
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 240 | 240 | 238
Participants
  Any drowsiness | 188 | 185 | 171
  Any irritability | 197 | 205 | 191
  Any loss of appetite | 135 | 127 | 112
  Any fever | 180 | 173 | 140

16. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE is any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of an AE regardless of intensity grade or relationship to study vaccination.
Time Frame: Within the 31-day (Days 0-30) follow up period after vaccination.
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 240 | 242 | 239
Participants | 153 | 165 | 159

17. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects. Any SAE = any SAE regardless of assessment of relationship to study vaccination.
Time Frame: During the entire study period (Month 0 to Month 3)
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 240 | 242 | 239
Participants | 9 | 5 | 4

ADVERSE EVENTS:
Time Frame: Solicited symptoms: 8-day follow-up period after vaccination; unsolicited AEs: 31-day follow-up period after vaccination; SAEs: during the entire study period (Months 0-3).
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Serious Adverse Events (participants affected / at risk) | 9/240 | 5/242 | 4/239
Other Adverse Events (participants affected / at risk) | 240/240 | 239/242 | 235/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK217744 Group 1 (N=240) | GSK217744 Group 2 (N=242) | Infanrix Hexa Group (N=239)
Bronchiolitis (Infections and infestations) | 4 | 0 | 3
Pneumonia (Infections and infestations) | 1 | 1 | 1
Amoebiasis (Infections and infestations) | 1 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Scaphocephaly (Congenital, familial and genetic disorders) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK217744 Group 1 (N=240) | GSK217744 Group 2 (N=242) | Infanrix Hexa Group (N=239)
Nasopharyngitis (Infections and infestations) | 53 | 64 | 51
Injection site induration (General disorders) | 22 | 14 | 25
Upper respiratory tract infection (Infections and infestations) | 14 | 21 | 15
Diarrhoea (Gastrointestinal disorders) | 13 | 13 | 21
Rhinitis (Infections and infestations) | 18 | 14 | 8
Conjunctivitis (Eye disorders) | 8 | 7 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 14 | 8
Pain (General disorders) | 190 | 183/240 | 155/238
Redness (General disorders) | 151 | 140/240 | 128/238
Swelling (General disorders) | 124 | 122/240 | 115/238
Drowsiness (General disorders) | 188 | 185/240 | 171/238
Irritability (General disorders) | 197 | 205/240 | 191/238
Loss of appetite (General disorders) | 135 | 127/240 | 112/238
Fever (General disorders) | 180 | 173 | 140

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.